CLINICAL TRIAL: NCT03818269
Title: Study of Subcutaneous Interstitial Pressure During Sepsis
Acronym: PISEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: DARGENT 2018
Record Dates: First submitted 2019-01-21; First posted 2019-01-28 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2021-09

CONDITIONS: Patients with Septic Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Septic shock (Other)
  Interventions: Procedure: Subcutaneous pressure measurement
- Control (Other)
  Interventions: Procedure: Subcutaneous pressure measurement

INTERVENTIONS:
Procedure: Subcutaneous pressure measurement — Subcutaneous interstitial measurement at D1 and D2

SUMMARY:
The pathophysiology of sepsis is characterized by the sudden onset of vasodilation and vascular permeability with capillary leakage. This leakage contributes to the development of generalized edema which is not clinically detectable below 4 litres but which becomes visible after a few days. The edema accumulates mainly at the subcutaneous level due to the high compliance of this tissue. Edema, and therefore hydrosodium overload, testifies to the severity of the inflammation. However, it could also be harmful in itself (affecting microcirculation and increasing mortality) as suggested by numerous clinical and experimental studies.

The transfer of fluids between vascular and interstitial compartments during sepsis therefore has a central role in the pathophysiology of the disease and associated mortality. These transfers are mainly controlled at the microvascular level (with constant permeability) by the difference between capillary (CP) and interstitial (IP) pressures. In healthy subjects, subcutaneous IP is discreetly negative (-1 mmHg) and varies very little. On the other hand, a sometimes drastic decrease in IP has been described in various localized and systemic inflammatory situations. These pressure variations may be explained by the collagen structure of the interstitial tissue and a change in the three-dimensional conformation of these macromolecules induced by inflammation mediators. In an animal model of sepsis, a study showed significantly lower pressure in a group of animals in endotoxic shock. IP has never been measured in humans during sepsis. The objective of this study is to analyze subcutaneous IP (SCIP) in patients with septic shock compared with controls in order to evaluate the direct role of interstitial tissue in the onset of edema during sepsis.

ELIGIBILITY:
Inclusion Criteria:

Criteria common to both groups:

* Adult,
* Admitted within the last 24 hours in intensive care,
* Under mechanical ventilation with orotracheal intubation,
* Without clinically detectable edema (in any area)
* Patient and/or guardian and/or close relative has given written consent

Patients included in the "septic shock" arm:

* Diagnosis of septic shock as defined by the "Sepsis-3" Consensus Conference (JAMA 2016) (34): documented or highly suspected infection with SOFA ≥ 2, persistent hypotension after correction of hypovolemia requiring vasopressor administration, and serum lactate > 2 mmol/l.
* Vascular filling < 50 ml/kg

Patients included in the control arm:

* Absence of sepsis and shock from any cause:

  * PAS > 100 mmHg
  * Absence of vasopressors
  * Preserved urine > 0.5 ml/kg/h
  * Normal serum lactate
* Crystalloid infusions < 50ml/kg over the previous 12 hours

Exclusion Criteria:

* not affiliated to national health insurance
* under court protection
* pregnant or breastfeeding
* Clinical disseminated intravascular coagulation (DIC) with hemorrhagic syndrome
* Admitted after resuscitation for cardiac arrest
* Presenting cardiogenic shock
* Presenting acute pancreatitis
* Severe overall dehydration (clinical signs of dehydration and natremia > 150mmol/l)
* Presenting metformin intoxication
* In severe sepsis or septic shock for more than 24 hours,
* Dying or for whom death seems imminent (within 24 hours),
* Hypersensitivity to lidocaine and/or prilocaine or local anesthetics of the amide type or to any of the excipients of EMLAPATCH®

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-26 (Actual); Primary Completion 2022-07-21 (Actual); Study Completion 2022-08-09 (Actual)

PRIMARY OUTCOMES:
Value of Initial subcutaneous interstitial pressure | Day 0
  Measure the difference between the subcutaneous interstitial pressure of patients in septic shock compared to patients without sepsis

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - CHU de DIJON, Dijon
  - HCL - Hôpital Edouard Herriot, Lyon

IPD SHARING:
Plan to Share IPD: No